CLINICAL TRIAL: NCT01979718
Title: The Post-operative Analgesia of the Virtual Reality Using a Mirror Therapy After Total Knee Arthroplasty: Prospective, Single-blind, Parallel Group, Randomized, Single Cohort Clinical Trial of Efficacy
Brief Title: The Post-operative Analgesia of the Virtual Reality Using a Mirror Therapy After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Associate Professor, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: chhwang3
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis, Knee; Nociceptive Pain; Virtual Reality
MeSH Terms: conditions — Osteoarthritis, Knee; Nociceptive Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Full term intervention (Experimental): * random selection
  * composed of the daily standard physical treatment and 1 session per one day over two weeks with a break on Saturday and Sunday (1 session is consisted of 50 repetitions of voluntary simultaneous flexion and extension of the both knees, taking a look at the mirrored virtual reality simulating the surgeried knee.
  Interventions: Device: Mirrored Virtual reality
- Half term intervention (Active Comparator): * random selection
  * composed of the daily standard physical treatment over two weeks and 1 session per one day over one weeks with a break on Saturday and Sunday (1 session is consisted of 50 repetitions of voluntary simultaneous flexion and extension of the both knees, taking a look at the mirrored virtual reality stimmulating the surgeried knee )
  Interventions: Device: Mirrored Virtual reality

INTERVENTIONS:
Device: Mirrored Virtual reality — Patients are required to look at the images of both lower extremities ranged from the perineal area to the foot. Virtual reality system records in real-time method both lower extremities. Following the validity assessement mirrored image of the surgeried lower extremity is re-formed using the virtusal reality system flipping the image of lower extremity not-surgeried and being calibration for the symmetricity.

SUMMARY:
It was well known that the mirror therapy could decrease pain of upper-limb amputated patients.

The mirror therapy is known to make a plastic change some parts of the brain perceiving the painful body part and modulating its signal by feedback of visual information mirrored with the corresponding contra-lateral normal parts.

In this study, post-operative analgesic efficiency of the virtual reality using a mirror therapy after total knee arthroplasty will be evaluated.

This clinical trial will be performed in the form of prospective, single-blind (i.e. assessor-blind), parallel group, randomized (allocation ratio 1:1), single cohort.

ELIGIBILITY:
Inclusion Criteria:

* patients who were transferred to RM after unilateral TKA

Exclusion Criteria:

* patients cannot freely move the contralat. leg d/t neurologic or musculoskeletal problems
* patients are not enough clear to indicate VAS
* patients cannot look at the virtual reality monitor d/t visual problem
* refusal of the participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | shortly after the 1st and 2nd session (5 days) intervention, and after 6 weeks after intervention
  The distance walked at a self-selected speed along a 40 cm corridor in 6 min. The distance was measured in meters, and more the meters better the result. A walking aid was used if needed.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) while resting | shortly after the 1st and 2nd session (5 days) intervention, and after 6 weeks after intervention
  checking the VAS while resting
Visual analogue scale (VAS) while moving | shortly after the 1st and 2nd session (5 days) intervention, and after 6 weeks after intervention
  checking the VAS while resting
Active ROM of flexion and extension on the knee | shortly after the 1st and 2nd session (5 days) intervention, and after 6 weeks after intervention
Tridol consumption per week | after the 1st and 2nd session (5 days) intervention
WOMAC index | shortly after the 1st and 2nd session (5 days) intervention, and after 6 weeks after intervention
Graded ambulation distances | shortly after the 1st and 2nd session (5 days) intervention, and after 6 weeks after intervention
  Grade 1: able to ambulate ≤5 feet Grade 2: able to ambulate >5 feet but <10 feet Grade 3: able to ambulate >10 feet but <30 feet Grade 4: able to ambulate ≥30 feet
Timed-stands test | shortly after the 1st and 2nd session (5 days) intervention, and after 6 weeks after intervention
  The patients were asked to rise from and sit down on a chair with a height of 45 cm, 10 times and as quickly as possible, without using the armrests. The time spent was recorded.
Side effects | after the 1st and 2nd session (5 days) intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Ph.D., Principal Investigator — Ulsan University Hospital; Sung Do Cho, M.D., Ph.D., Principal Investigator — Ulsan University Hospital; Youngjoon Chee, Ph.D., Principal Investigator — Department of Biomedical Engineering, University of Ulsan; Kyo-In Koo, Ph.D., Principal Investigator — Department of Biomedical Engineering, University of Ulsan
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided